CLINICAL TRIAL: NCT03927664
Title: Conception and Validation of a Clinico-radiological Classification of Peritoneal Tuberculosis
Brief Title: Clinico-radiological Classification of Peritoneal Tuberculosis
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vishal Sharma, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/5243/Study/019
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Tuberculosis; Tuberculosis; Abdomen (Etiology); Tuberculosis, Peritoneal
MeSH Terms: conditions — Tuberculosis; Peritonitis, Tuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peritoneal Tuberculosis: Patients diagnosed with peritoneal tuberculosis and who have undergone a computed tomographic examination
  Interventions: Other: Radiological assessment

INTERVENTIONS:
Other: Radiological assessment — Radiological assessment of findings in the peritoneum, omentum, mesentery, ascites and other abdominal findings

SUMMARY:
Traditionally, peritoneal tuberculosis has been classified as wet-ascitic, dry-plastic type and fibrotic -fixed types. there is substantial overlap between these definitions and the clinical implication of the categorisation into the three patterns is unclear.

The clinical presentation will be used to divide participants into 1) Abdominal distension dominant disease or 2) Pain Dominant and/or 3) Obstruction dominant peritoneal tuberculosis. The radiological findings between these groups will be compared if findings on radiology are discriminative of these three patterns of presentation.

DETAILED DESCRIPTION:
The study will be conducted as two parts

1. Derivation group:

   Screening population: Patients with abdominal tuberculosis treated in the gastroenterology unit from Jan 2017-Dec 2018 This will involve a retrospective study where the patients who have been treated for peritoneal tuberculosis and have full records available (as hospital records or Gut-Tuberculosis clinic files) will be included and their clinical details and radiological findings (from CT films or images) will be entered and compared. The radiological findings between these groups will be compared if findings on radiology are discriminative of these three patterns of presentation.
2. Validation Study: This will include prospective study of patients who have underwent computed tomography for evaluation of abdominal complaints and are eventually diagnosed to have peritoneal tuberculosis. The radiological parameters derived from the derivation group will be tested to predict the clinical presentation.

At the end of the study,the feasibility of a clinico-radiological classification of peritoneal tuberculosis.

The clinical details will be recorded and will include demographic details, diagnostic work-up (confirmed/probable), follow-up and classification into one of the three patterns of presentation

1. Distension dominant: Presence of abdominal distention or discomfort, Lack of pain
2. Pain dominant: Patients having associated significant abdominal pain necessitating analgesics or interfering with routine activities
3. Obstruction dominant; Clear historical and/or radiological evidence of intestinal obstruction like abdominal pain associated with distension and obstipation

Computed tomographic scans/images will be assessed by the two radiologists separately and resolved by consensus The radiologists will not have access to any clinical details The findings will be recorded on a proforma and will include determination of presence and extent of ascites, loculated ascites, peritoneal nodules or masses, omental involvement as nodules or masses, mesenteric adenopathy, masses, abdominal lymphadenopathy, presence of clumped loops, adhesions, abdominal cocoon etc The three groups will be compared for these radiological patterns and a possible correlation between any radiological findings and the clinical presentation will be derived.

The classification derived from the derivation cohort will be tested in validation cohort which will be a prospective study. The clinical presentation will be recorded. The CT scans will be reviewed by two radiologists blinded to clinical details and the clinical presentation will be compared with categorisation based on the radiological findings.

ELIGIBILITY:
Inclusion Criteria

* Patients diagnosed with peritoneal tuberculosis
* Patients who have undergone a computed tomographic examination

Exclusion Criteria:

* Age < 12
* Unclear diagnosis
* More than one etiology for ascites
* Not willing for consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with peritoneal tuberculosis or being treated as peritoneal tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Correlation of radiological characterization of classification with clinical presentation | 3 months of diagnosis
  Clinical presentation will be classified as 1) Distension dominant 2) Pain dominant 3) Obstruction dominant This will be correlated with the categorisation based on radiologic findings and correlation between the radiological category an actual clinical category will be studied

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Sharma, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (2):
- India (2):
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Department of Gastroenterology, Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahamed Z R, Shah J, Agarwala R, Kumar-M P, Mandavdhare HS, Gupta P, Singh H, Sharma A, Dutta U, Sharma V. Controversies in classification of peritoneal tuberculosis and a proposal for clinico-radiological classification. Expert Rev Anti Infect Ther. 2019 Aug;17(8):547-555. doi: 10.1080/14787210.2019.1642746. Epub 2019 Jul 17. PMID 31293195